CLINICAL TRIAL: NCT04717856
Title: Evaluation of the Use of the GenXpert to Detect Hepatitis C RNA Using a Finger Prick; a Cross-sectional, Multicentre Study Among Drug Users
Brief Title: Evaluation of the Use of the GenXpert to Detect Hepatitis C RNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CEPHEID-01
Record Dates: First submitted 2020-11-26; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Drug Use; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- drug users (Other)
  Interventions: Other: screening: HCV RNA test and risk factors questionaire

INTERVENTIONS:
Other: screening: HCV RNA test and risk factors questionaire — Screening by using a rapid finger prick test for HCV RNA and a questionnaire to assess risk factors.

SUMMARY:
The results of the GX device are equivalent to standard venous blood sampling. With this study we are going to determine the prevalence in drug users with difficult venous access. On the other hand, we want to look at the place this device can have in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Have recently or ever used drugs
* Older than 18 years
* Written informed consent

Exclusion Criteria:

* Not being able to speak the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-10-21 (Estimated); Study Completion 2021-10-21 (Estimated)

PRIMARY OUTCOMES:
Questionaire to determine the satisfaction of the use of the GenXpert | baseline
  1. To determine how the caregiver and the client experience the use of the GenXpert and what place the device can have in primary care. a. A questionnaire to determine the satisfaction of the user and the person tested

SECONDARY OUTCOMES:
The detection of HCV RNA | Baseline
  a. One finger prick to measure the HCV RNA. These blood samples are processed directly using the HCV Viral Load fingerstick cartridge which is processed via the GenXpert device.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University, Diepenbeek, Belgium